CLINICAL TRIAL: NCT01606878
Title: A Phase 1 Study of Crizotinib in Combination With Conventional Chemotherapy for Relapsed or Refractory Solid Tumors or Anaplastic Large Cell Lymphoma
Brief Title: Crizotinib and Combination Chemotherapy in Treating Younger Patients With Relapsed or Refractory Solid Tumors or Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1212; NCI-2012-01968 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000734059; ADVL1212; ADVL1212 (Other: COG Phase I Consortium); ADVL1212 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Childhood Solid Neoplasm; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Neuroblastoma
Keywords: Crizotinib; Chemotherapy; Solid Tumors; Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Neuroblastoma | interventions — Crizotinib; Cyclophosphamide; Dexrazoxane; Razoxane; Doxorubicin; Topotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A (crizotinib, cyclophosphamide, topotecan hydrochloride) (Experimental): Patients receive crizotinib (oral solution) PO BID on days 1-21, cyclophosphamide IV QD on days 1-5, and topotecan hydrochloride IV QD on days 1-5. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
  Interventions: Drug: Crizotinib; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration; Drug: Topotecan Hydrochloride
- Part B (crizotinib, vincristine, dexrazoxane, doxorubicin) (Experimental): Patients receive crizotinib (oral solution) PO BID as in Part A. Patients also receive vincristine sulfate IV on day 1, dexrazoxane hydrochloride IV on day 1, and doxorubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
  Interventions: Drug: Crizotinib; Drug: Dexrazoxane Hydrochloride; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Part C (crizotinib, cyclophosphamide, topotecan hydrochloride) (Experimental): Patients receive crizotinib (capsule formulation) PO BID, cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration; Drug: Topotecan Hydrochloride
- Part D (crizotinib, cyclophosphamide, topotecan hydrochloride) (Experimental): Patients receive crizotinib (microsphere formulation) PO BID, cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Drug: Crizotinib — Given PO
  Other Names: MET Tyrosine Kinase Inhibitor PF-02341066; PF-02341066; PF-2341066; Xalkori
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Part A (crizotinib, cyclophosphamide, topotecan hydrochloride); Part C (crizotinib, cyclophosphamide, topotecan hydrochloride); Part D (crizotinib, cyclophosphamide, topotecan hydrochloride)
Drug: Dexrazoxane Hydrochloride — Given IV
  Other Names: Cardioxane; Totect; Zinecard
  Arms: Part B (crizotinib, vincristine, dexrazoxane, doxorubicin)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Part B (crizotinib, vincristine, dexrazoxane, doxorubicin)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Part A (crizotinib, cyclophosphamide, topotecan hydrochloride); Part C (crizotinib, cyclophosphamide, topotecan hydrochloride); Part D (crizotinib, cyclophosphamide, topotecan hydrochloride)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Part B (crizotinib, vincristine, dexrazoxane, doxorubicin)

SUMMARY:
This phase I trial studies the side effects and the best dose of crizotinib when given together with combination chemotherapy in treating younger patients with solid tumors or anaplastic large cell lymphoma that has returned or does not respond to treatment. Crizotinib may stop the growth of tumor or cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, topotecan hydrochloride, dexrazoxane hydrochloride, doxorubicin hydrochloride, and vincristine sulfate, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving crizotinib together with combination chemotherapy may be a better treatment for patients with solid tumors or anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD) of crizotinib administered orally twice daily in combination with topotecan (topotecan hydrochloride) and cyclophosphamide in children with refractory/relapsed solid tumors or anaplastic large cell lymphoma (ALCL).

II. To define and describe the toxicities of crizotinib in combination with topotecan and cyclophosphamide administered on this schedule.

III. To estimate the recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD) of crizotinib administered orally twice daily in combination with vincristine (vincristine sulfate) and doxorubicin (doxorubicin hydrochloride)/dexrazoxane (dexrazoxane hydrochloride) in children with refractory/relapsed solid tumors or ALCL.

IV. To define and describe the toxicities of crizotinib in combination with vincristine and doxorubicin/dexrazoxane administered on this schedule.

V. To characterize the pharmacokinetics of crizotinib in children with relapsed/refractory cancer when combined with either topotecan and cyclophosphamide or vincristine and doxorubicin/dexrazoxane.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of crizotinib in combination with either topotecan and cyclophosphamide or vincristine and doxorubicin/dexrazoxane within the confines of a Phase 1 study.

II. To preliminarily examine the relationship between anaplastic lymphoma kinase (ALK) status in patients with neuroblastoma or ALCL and response to crizotinib in combination with either topotecan and cyclophosphamide or vincristine and doxorubicin/dexrazoxane.

III. To preliminarily examine the relationship between minimal residual disease (MRD) status and clinical response to crizotinib in combination with either topotecan and cyclophosphamide or vincristine and doxorubicin/dexrazoxane in patients with ALCL.

IV. To use a questionnaire to gather preliminary information on the palatability of the oral solution formulation of crizotinib.

V. To examine ALK and MET proto-oncogene (c-Met) expression, copy number and mutations status in archival tumor tissue from solid tumor and ALCL patients.

VI. To use a questionnaire to gather information on the acceptability of the crizotinib capsule formulation.

OUTLINE: This is a dose-escalation study of crizotinib. Patients are assigned to Part A or Part B based on the treating physician's choice and availability of a reservation. After closure of Part A and Part B, patients are assigned to Part C.

PART A (CLOSED TO ACCRUAL 10/3/14): Patients receive crizotinib (oral solution) orally (PO) twice daily (BID) on days 1-21, cyclophosphamide intravenously (IV) once daily (QD) on days 1-5, and topotecan hydrochloride IV QD on days 1-5. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

PART B (CLOSED TO ACCRUAL 10/3/14): Patients receive crizotinib (oral solution) PO BID as in Part A. Patients also receive vincristine sulfate IV on day 1, dexrazoxane hydrochloride IV on day 1, and doxorubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

PART C: Patients receive crizotinib (capsule formulation) PO BID, cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

PART D: Patients receive crizotinib (microsphere formulation) PO BID, cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of malignancy at original diagnosis or relapse; all patients with relapsed or refractory solid tumors or anaplastic large cell lymphoma (ALCL) are eligible except for patients with primary or metastatic central nervous system (CNS) tumors or patients with primary cutaneous ALCL
* Patients must have either measurable or evaluable disease
* Patients current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 60% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy

  * Myelosuppressive chemotherapy:

    * Solid tumors: at least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
    * ALCL:

      * Patients with ALCL who relapse while receiving standard maintenance chemotherapy will not be required to have a waiting period before enrollment onto this study
      * Patients who relapse while they are not receiving standard maintenance therapy, must have fully recovered from all acute toxic effects of prior therapy; at least 14 days must have elapsed after the completion of cytotoxic therapy
  * Hematopoietic growth factors: at least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Biologic (anti-neoplastic agent): at least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Immunotherapy: at least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Monoclonal antibodies: at least 3 half-lives of the antibody after the last dose of a monoclonal antibody
  * Radiation therapy (XRT):

    * Solid tumors: at least 14 days after local palliative XRT (small port); >= 6 weeks must have elapsed since treatment with therapeutic doses of metaiodobenzylguanidine (MIBG); at least 150 days must have elapsed if prior total body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow (BM) radiation
    * ALCL: at least 14 days after local palliative XRT (small port); at least 84 days must have elapsed if prior TBI, craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial BM radiation
  * Stem cell infusion without TBI: no evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant and >= 42 days for autologous stem cell infusion after iodine (I)131-MIBG therapy
  * Patients must not have received prior therapy with crizotinib
  * Prior anthracycline dose: patients with a total lifetime cumulative anthracycline dose of > 650 mg/m^2 at the time of enrollment are not eligible for Part B of the study
* For patients with solid tumors or ALCL without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years: 0.6 mg/dL
  * Age 2 to < 6 years: 0.8 mg/dL
  * Age 6 to < 10 years: 1 mg/dL
  * Age 10 to < 13 years: 1.2 mg/dL
  * Age 13 to < 16 years: 1.5 mg/dL (males) and 1.4 mg/dL (females)
  * Age >= 16 years: 1.7 mg/dL (males) and 1.4 mg/dL (females)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Corrected QT interval (QTc) =< 480 msec
* For patients on Part B: shortening fraction of >= 27% by echocardiogram or ejection fraction of >= 50% by gated radionuclide study
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Part C: Patients must have a body surface area (BSA) >= 1.07 m^2 at the time of study enrollment
* Part D: Patients must have a body surface area (BSA) >= 0.43 m^2 at the time of study enrollment
* Tumor tissue must be sent; if tumor tissue is unavailable, the study chair must be notified prior to enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during treatment and for 3 months after stopping treatment
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients chronically receiving medications known to be metabolized by cytochrome P 450, family 3, subfamily A, polypeptide 4 (CYP3A4) and with narrow therapeutic indices including pimozide, aripiprazole, triazolam, ergotamine and halofantrine are not eligible; the topical use of these medications (if applicable) is allowed
* Patients chronically receiving drugs that are known potent CYP3A4 inhibitors within 7 days prior to study enrollment, including but not limited to ketoconazole, itraconazole, miconazole, clarithromycin, erythromycin, ritonavir, indinavir, nelfinavir, saquinavir, amprenavir, delavirdine, nefazodone, diltiazem, verapamil, and grapefruit juice are not eligible; the topical use of these medications (if applicable), e.g. 2% ketoconazole cream, is allowed
* Patients chronically receiving drugs that are known potent CYP3A4 inducers within 12 days prior to study enrollment, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, tipranavir, ritonavir, and St. John?s wort are not eligible; the topical use of these medications (if applicable) is allowed
* Patients receiving PPIs and H2 blockers are not eligible for Part D
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who have a primary or metastatic CNS tumor at the time of study enrollment are not eligible; a prior history of metastatic CNS tumor is allowed as long as there is no evidence of CNS disease at study enrollment
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Parts A and B: Patients who are able to swallow liquid or use a nasogastric or gastrostomy (G) tube are eligible
* Part C: Patients must be able to swallow intact capsules
* Part D: Patients must be able to swallow liquid

Ages: 13 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Greengard, Principal Investigator — COG Phase I Consortium
Locations (23):
- United States (22):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Greengard E, Mosse YP, Liu X, Minard CG, Reid JM, Voss S, Wilner K, Fox E, Balis F, Blaney SM, Adamson PC, Weigel BJ. Safety, tolerability and pharmacokinetics of crizotinib in combination with cytotoxic chemotherapy for pediatric patients with refractory solid tumors or anaplastic large cell lymphoma (ALCL): a Children's Oncology Group phase 1 consortium study (ADVL1212). Cancer Chemother Pharmacol. 2020 Dec;86(6):829-840. doi: 10.1007/s00280-020-04171-4. Epub 2020 Oct 23. PMID 33095287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a dose-escalation study of crizotinib. Patients are assigned to Part A or Part B based on the treating physician's choice and availability of a reservation. After closure of Part A and Part B, patients are assigned to Part C and Part D.
Groups:
- Part A Dose Level 1: Patients receive 165 mg/m^2 crizotinib (oral solution) PO BID on days 1-21, 250 mg/m^2 cyclophosphamide IV QD on days 1-5, and topotecan hydrochloride IV QD on days 1-5. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
- Part A Dose Level 2: Patients receive 215 mg/m^2 crizotinib (oral solution) PO BID on days 1-21, 250 mg/m^2 cyclophosphamide IV QD on days 1-5, and topotecan hydrochloride IV QD on days 1-5. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
- Part B Dose Level 1: Patients receive 165 mg/m^2 crizotinib (oral solution) PO BID as in Part A. Patients also receive 1.5 mg/m^2 vincristine sulfate IV on day 1, 450 mg/m^2 dexrazoxane hydrochloride IV on day 1, and 45 mg/m^2 doxorubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
- Part B Dose Level 2: Patients receive 215 mg/m^2 crizotinib (oral solution) PO BID as in Part A. Patients also receive 1.5 mg/m^2 vincristine sulfate IV on day 1, 450 mg/m^2 dexrazoxane hydrochloride IV on day 1, and 45 mg/m^2 doxorubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
- Part B Dose Level 3: Patients receive 280 mg/m^2 crizotinib (oral solution) PO BID as in Part A. Patients also receive 1.5 mg/m^2 vincristine sulfate IV on day 1, 450 mg/m^2 dexrazoxane hydrochloride IV on day 1, and 45 mg/m^2 doxorubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/3/14)
- Part C Dose Level 1: Patients receive 165 mg/m^2 crizotinib (capsule formulation) PO BID, 250 mg/m^2 cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
- Part C Dose Level 2: Patients receive 215 mg/m^2 crizotinib (capsule formulation) PO BID, 250 mg/m^2 cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
- Part C Dose Level 3: Patients receive 280 mg/m^2 crizotinib (capsule formulation) PO BID, 250 mg/m^2 cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
- Part D Dose Level 1: Patients receive 165 mg/m^2 crizotinib (microsphere formulation) PO BID, 250 mg/m^2 cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
- Part D Dose Level 2; Part PK Dose Level 2: Patients receive 215 mg/m^2 crizotinib (microsphere formulation) PO BID, 250 mg/m^2 cyclophosphamide IV QD, and topotecan hydrochloride IV QD as in Part A. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Started | 6 | 4 | 5 | 3 | 3 | 4 | 6 | 3 | 6 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 4 | 5 | 3 | 3 | 4 | 6 | 3 | 6 | 3 | 3
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 2 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2 | Total
Number analyzed (Participants) | 6 | 4 | 5 | 3 | 3 | 4 | 6 | 3 | 6 | 3 | 3 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 2 | 2 | 3 | 2 | 5 | 3 | 6 | 3 | 1 | 35
  Between 18 and 65 years | 2 | 0 | 3 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [4.0 to 21.0] | 12.5 [7.0 to 17.0] | 19 [7.0 to 21.0] | 6 [6.0 to 19.0] | 11 [10.0 to 17.0] | 17.5 [15.0 to 20.0] | 15 [9.0 to 20.0] | 17 [13.0 to 17.0] | 13.5 [1.0 to 17.0] | 17 [10.0 to 18.0] | 20 [11.0 to 21.0] | 15 [1.0 to 21.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 2 | 3 | 1 | 3 | 1 | 2 | 22
  Male | 4 | 1 | 3 | 2 | 1 | 2 | 3 | 2 | 3 | 2 | 1 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 7
  Not Hispanic or Latino | 6 | 4 | 4 | 2 | 2 | 4 | 4 | 3 | 5 | 3 | 2 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 9
  White | 3 | 3 | 4 | 3 | 2 | 3 | 5 | 2 | 4 | 3 | 3 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Crizotinib
Description: The MTD of crizotinib administered with combination chemotherapy based on the incidence of dose-limiting toxicity (DLT) at which fewer than one-third of patients experience DLT, as assessed by NCI CTCAE version 4.0.
Time Frame: Up to 21 days
Population: Parts A, B and D MTD/RP2D were not assessed. As of Amendment #3, due to the possibility that many of the non-hematologic DLTs observed to date on the study are related to the palatability of the OS rather than due to true toxicity of the investigational agent, Parts A and B were closed and Part C was then opened to determine the MTD/ RP2D. As of Amendment #4, a new microsphere formulation was added for Part D, but there was no MTD/RP2D.
Measure: Number; unit: mg/m^2
Arm/Group | Part C (Crizotinib, Cyclophosphamide, Topotecan Hydrochloride)
Number analyzed (Participants) | 11
mg/m^2 | 215

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT)
Description: Number of patients of all DLT reported as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. stratified by dose level and study part.
Time Frame: Up to 21 days
Population: All Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 3 | 3
Participants | 2 | 2 | 0 | 0 | 2 | 0 | 1 | 2 | 3 | 3 | 1

3. Primary Outcome: Area Under the Concentration
Description: Median (min, max) of the area under the concentration time curve for crizotinib assessed in course 1 at 1, 2, 4, 6-8 hours, and 15-21 days post-administration stratified by dose level and study part.
Time Frame: Up to 21 days
Population: All Toxicity evaluable patients. There were no data for Part A Dose Level 2, Part B Dose Level 3, and Part D Dose Level 1.
Measure: Median (Full Range); unit: hr*ug/mL
Arm/Group | Part A Dose Level 1 | Part B Dose Level 1 | Part B Dose Level 2 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 5 | 3 | 3 | 1 | 5 | 1 | 2 | 2
hr*ug/mL | 3792.5 [1808.8 to 5520.3] | 1549.3 [811.4 to 2544.3] | 4070.5 [3588.0 to 10145.9] | 1612 [1612.0 to 1612.0] | 3796.6 [2976.0 to 7299.3] | 7462.8 [7462.8 to 7462.8] | 3248 [3109.9 to 3386.1] | 8881.3 [5701.6 to 12061.0]

4. Secondary Outcome: Response Rate
Description: Number of patients of response-evaluable participants with response (CR/PR) assessed according to Response Evaluation Criteria in Solid Tumors version 1.1 including CR: disappearance of all target and non-target lesions; PR: at least 30% decrease in the sum of the diameters of target lesions
Time Frame: Up to 2 years
Population: Evaluable patients for response
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 6 | 4 | 5 | 3 | 3 | 4 | 6 | 3 | 6 | 3 | 3
Participants | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0

5. Secondary Outcome: ALK Status and Response to Crizotinib
Description: Number of patients who respond (CR/PR) to crizotinib in combination with either topotecan and cyclophosphamide or vincristine and doxorubicin/dexraroxane stratified by ALK positive or negative status
Time Frame: up to 2 years
Population: Neuroblastoma patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants
  ALK Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALK Negative | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: MRD Status and Response to Crizotinib
Description: Frequency (%) of patients who respond (CR/PR) to crizotinib in combination with either topotecan and cyclophosphamide or vincristine and doxorubicin/dexraroxane stratified by MRD status
Time Frame: Up to 2 years
Population: Outcome Measure was specific to ALCL patients. There were zero ALCL patients, therefore, there are no data to report.
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: ALK Expression for Crizotinib
Description: Median (p25, p75) ALK expression stratified by dose level and study part
Time Frame: Up to 7 days
Population: ALK expression data were not and never will be collected.
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Acceptability of Crizotinib Capsule Formulation Palatability
Description: Number of patients who at least accept palatability of capsule formulation in the first week
Time Frame: Up to 1 week
Population: All Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 3 | 0 | 0 | 3

9. Secondary Outcome: Acceptability of Crizotinib Microsphere Formulation Palatability
Description: Number of patients who at least accept palatability of microsphere formation in the first week
Time Frame: Up to 1 week
Population: All Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study.
  Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Part A Dose Level 1 | Part A Dose Level 2 | Part B Dose Level 1 | Part B Dose Level 2 | Part B Dose Level 3 | Part C Dose Level 1 | Part C Dose Level 2 | Part C Dose Level 3 | Part D Dose Level 1 | Part D Dose Level 2 | Part PK Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 1/5 | 0/3 | 0/3 | 1/4 | 0/6 | 0/3 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/4 | 1/5 | 1/3 | 2/3 | 3/4 | 3/6 | 1/3 | 3/6 | 3/3 | 2/3
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 5/5 | 3/3 | 3/3 | 4/4 | 6/6 | 3/3 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1 (N=6) | Part A Dose Level 2 (N=4) | Part B Dose Level 1 (N=5) | Part B Dose Level 2 (N=3) | Part B Dose Level 3 (N=3) | Part C Dose Level 1 (N=4) | Part C Dose Level 2 (N=6) | Part C Dose Level 3 (N=3) | Part D Dose Level 1 (N=6) | Part D Dose Level 2 (N=3) | Part PK Dose Level 2 (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1 (N=6) | Part A Dose Level 2 (N=4) | Part B Dose Level 1 (N=5) | Part B Dose Level 2 (N=3) | Part B Dose Level 3 (N=3) | Part C Dose Level 1 (N=4) | Part C Dose Level 2 (N=6) | Part C Dose Level 3 (N=3) | Part D Dose Level 1 (N=6) | Part D Dose Level 2 (N=3) | Part PK Dose Level 2 (N=3)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 2 | 2 | 2 | 2 | 4 | 1 | 4 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3 | 4 | 3 | 3 | 1 | 5 | 2 | 6 | 2 | 2
Alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 3 | 0 | 4 | 6 | 0 | 3 | 2 | 0
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 4 | 5 | 3 | 3 | 4 | 6 | 3 | 6 | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 2 | 5 | 2 | 3 | 1 | 4 | 3 | 4 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 2 | 2 | 3 | 1 | 5 | 2 | 4 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 1 | 1 | 3 | 5 | 2 | 3 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, CERVICAL ADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, ECCHYMOSES ON BILATERAL EXTREMITIES (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 1 | 2 | 2 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Cardiac disorders - Other, INCOMPLETE RIGHT BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac disorders - Other, LEFT VENTRICULAR HYPERTOPHY (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 2 | 2 | 2 | 0 | 4 | 1 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 2 | 1 | 3 | 4 | 2 | 3 | 2 | 0
Creatinine increased (Investigations) | 2 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 4 | 3 | 2 | 2 | 2 | 4 | 2 | 3 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 3 | 4 | 0 | 1 | 1 | 1
Ear and labyrinth disorders - Other, ERYTHEMA - OUTER EAR (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Edema face (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Endocrine disorders - Other, VITAMIN D DEFICIENCY (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, "GHOST"APPEARANCE OF VISION. (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, 20/160 VISION IN RIGHT EYE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, BLACK SPOTS/FLOATERS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, CALCIFICATIONS IN BILAT GLOBES FROM PRIOR RETINOBLASTOMA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, CHANGES IN LOW LIGHT (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, CLEAR DRAINAGE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, CRUSTY EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, DECREASED VISUAL ACUITY (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, DOUBLE VISION (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, EYELID SWELLING (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, GHOSTLY/SHADOWING/3D VISION (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, ITCHY EYES (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, LIGHT PERCEPTION IN LEFT EYE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, NEARSIGHTEDNESS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, PURPLE EYELIDS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, SEEING AURA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, SEEING BARS IN HIS VISION (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, SEEING STREAKS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, STREAKING (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, TRACERS (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, TRAILING VISION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, TRICHIASIS (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, TWITCHING OF HER EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, VISUAL DISTURBANCE (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, VISUAL IMPAIRMENT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, VISUAL STREAKING (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 4 | 3 | 3 | 2 | 2 | 4 | 6 | 3 | 5 | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 1 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 4 | 2 | 0 | 2 | 0 | 3 | 3 | 2 | 3 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
GGT increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorders - Other, CHIPPED TOOTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, FOAMY SALIVA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, HEARTBURN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, LIP SORE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, TOOTH PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, WISDOM TOOTH ERUPRTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, BLEEDING GUMS (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 1 | 1 | 0 | 1 | 4 | 2 | 2 | 3 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hematuria (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disorders - Other, HEPATOSPLENOMEGALY (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 0 | 2 | 3 | 2 | 2 | 3 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 2 | 1 | 0 | 3 | 2 | 1 | 1 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 2 | 6 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 4 | 3 | 1 | 2 | 3 | 4 | 3 | 2 | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2 | 1 | 2 | 5 | 0 | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3 | 2 | 1 | 1 | 4 | 3 | 2 | 3 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 1 | 1 | 2 | 4 | 1 | 3 | 2 | 3
Hypotension (Vascular disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 3 | 2 | 1
Hypothyroidism (Endocrine disorders) | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
INR increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Immune system disorders - Other, ALLERGY TO ONDANSETRON (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune system disorders - Other, IMMUNOCOMPROMISED (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, CANDIDA (G-TUBE SITE) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, COLD SORE (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, E. COLI (BOTH CVL LUMENS) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, HSV-1 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, LOWER RESPIRATORY INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, PSEUDOMONAS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, PULMONARY (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, RHINOVIRUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, THRUSH (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, ABRASION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, BLEEDING LOVENOX INJECTION SITES (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, IRRITATED THROAT FROM INTUBATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury, poisoning and procedural complications - Other, MILD SCALP SWELLING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 1
Investigations - Other, ALK PHOS DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ANION GAP INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, BUN DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BUN INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BUN, DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, CHLORIDE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, CREATININE DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, CRP, INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, DECREASED BUN (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, DECREASED SERUM PROTEIN (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, DECREASED TOTAL SERUM PROTEIN (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED CRP (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, HYPERAMMONEMIA (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, INCREASED CHLORIDE (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, INR DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, LACTATE INCREASED - CAP BLOOD GAS (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, NON FASTING HYPERGLYCEMIA (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, NON-FASTING GLUCOSE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, PHOSPHATE INCREASE (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, SERUM PROTEIN DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TOTAL PROTEIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 6 | 4 | 5 | 3 | 3 | 4 | 6 | 3 | 6 | 3 | 2
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, INCREASED PHOSPHOROUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, NON FASTING GLUCOSE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolism and nutrition disorders - Other, TOTAL PROTEIN DECREASED (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, COLD EXTREMITIES (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, INABILITY TO OPEN MOUTH WELL (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, LIMITED ROM D/T PAIN FROM NECK MASS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, MUSCLE STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 4 | 5 | 3 | 3 | 3 | 6 | 3 | 5 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, ALTERED MENTAL STATUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, HORNER'S SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 6 | 4 | 3 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 0 | 1 | 3 | 2 | 1 | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 6 | 4 | 5 | 2 | 3 | 3 | 6 | 2 | 6 | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Psychiatric disorders - Other, ADHD (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, EMOTIONAL (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Renal and urinary disorders - Other, DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, FANCONI SYNDROME (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, GLUCOSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, KETONURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, SIADH (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, TRACE KETONES (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Reproductive system and breast disorders - Other, HYPOVENTILATION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, CRACKLES IN RIGHT LUNG (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, DIMINISHED AIR ENTRY IN LUNG (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, NASAL DISCHARGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 5 | 0 | 1 | 1 | 0 | 2 | 4 | 2 | 4 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, ABRASION ON CHIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, BULLOUS LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, CRADLE CAP (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, DIAPER RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA AROUND FINGERNAILS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA AT G-TUBE SITE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMATOUS EYELIDS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, INFLAMED RIGHT INDEX FINGER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, INSECT BITES (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PURPLE COLOR TO HANDS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, RED, FLAT RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, SKIN ABRASION ANKLE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, EGD (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Unequal limb length (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular disorders - Other, AV THROMBUS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vascular disorders - Other, CHRONIC OCCLUSION OF THE SUBCLAVIAN AND BRACHIOCEPHLIC VEINS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4 | 5 | 3 | 3 | 4 | 5 | 3 | 6 | 3 | 3
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 3 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 6 | 4 | 5 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT01606878/Prot_SAP_000.pdf